CLINICAL TRIAL: NCT04710134
Title: Efficacy of Reslizumab Dose Escalation in Patients With Severe Asthma and Persistent Sputum Eosinophilia Despite Standard Dose Therapy
Brief Title: Efficacy of Reslizumab Dose Escalation in Patients With Severe Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Teva Canada (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RES-2020-20
Record Dates: First submitted 2021-01-08; First posted 2021-01-14 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Asthma; Eosinophilic
Keywords: Asthma; Eosinophilic bronchitis; Reslizumab
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma | interventions — reslizumab

STUDY DESIGN:
Intervention Model Description: Patients will initially all receive 3 mg/kg of reslizumab. After 16 weeks of treatment, those patients that have uncontrolled sputum eosinophilia will be escalated to 4 mg/kg; the remaining patients will continue on 3 mg/kg. After a further 16 weeks of therapy, those that still have uncontrolled sputum eosinophilia will receive 5 mg/kg; the remaining patients will continue on the dose they were receiving (i.e., either 3 or 4 mg/kg).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Reslizumab 3 mg/kg (Active Comparator): All patients will initially receive reslizumab 3 mg/kg for at least 16 weeks.
  Interventions: Biological: Reslizumab
- Reslizumab 4 mg/kg (Active Comparator): Patients who have uncontrolled sputum eosinophilia at 16 weeks will receive an increased dose of 4 mg/kg for the next 16 weeks. The patients with controlled eosinophilia will continue to receive 3 mg/kg.
  Interventions: Biological: Reslizumab
- Reslizumab 5 mg/kg (Active Comparator): Patients who have uncontrolled sputum eosinophilia who were previously receiving reslizumab at 4 mg/kg at 32 weeks will receive an increased dose of 5 mg/kg for the next 16 weeks. The patients remaining patients will continue on the dose they were receiving (i.e., either 3 mg/kg or 4 mg/kg).
  Interventions: Biological: Reslizumab

INTERVENTIONS:
Biological: Reslizumab — Reslizumab 3,4, or 5 mg/kg IV q4 weeks

SUMMARY:
Dose escalation of reslizumab can ameliorate sputum eosinophilia in severe asthmatics who have persistent sputum eosinophilia despite treatment with reslizumab at the standard dose.

DETAILED DESCRIPTION:
Monoclonal antibody therapies targeting the interleukin-5 (IL-5) pathway, critical for maintaining eosinophil homeostasis, have been developed as adjunct therapy for severe asthma with an eosinophilic phenotype. Reslizumab/Cinqair is an approved/marketed product administered monthly by intravenous to severe eosinophilic asthmatics at 3mg/kg. However some patients do exhibit sputum eosinophilia at this dosage. We are investigating whether those that receive 3mg/kg that have persistent sputum eosinophils would benefit at a higher dose of 4mg/kg and those that still exhibit sputum eosinophils at this elevated dose would show improvement at 5mg/kg.

The overall aim of this study is to determine whether dose escalation of reslizumab can ameliorate sputum eosinophilia in severe asthmatics who have persistent sputum eosinophilia despite treatment with reslizumab at the standard dose.

ELIGIBILITY:
Inclusion Criteria:

1. Asthma confirmed within the past 2 years by:

   a. A ≥12% improvement in forced expiratory volume in 1 second (FEV1) after use of a beta agonist, or a methacholine challenge test showing a ≥20% reduction in FEV1 after a concentration of ≤8 mg/mL of methacholine
2. Blood eosinophils ≥400 cells/µL and/or sputum eosinophils ≥3% (or presence of moderate-to-many free eosinophil granules) at the time of study enrollment
3. Treated with an inhaled corticosteroid at a dose of ≥1500 µg of fluticasone propionate (or equivalent) and a long-acting beta agonist with or without oral corticosteroids
4. Ability to provide informed consent

Exclusion Criteria:

1. Current smokers, ex-smokers with greater than 20 pack-year history or ex-smokers who have smoked within the past 6 months
2. Any comorbidity that the investigator believes is a contraindication including but not limited to any respiratory (e.g., chronic obstructive pulmonary disease, allergic bronchopulmonary aspergillosis, pulmonary fibrosis), cardiovascular (e.g., congestive cardiac failure, pulmonary hypertension), hematological, gastrointestinal, immunological, musculoskeletal, infectious, or neoplastic disease
3. Currently treated with another biologic agent (excluding denosumab for osteoporosis)
4. Use of anti-IL-5 (other than reslizumab) or anti-IgE mAb use within the past one month
5. Use of a systemic immunosuppressive or immunomodulatory agent within 6 months prior to study entry
6. Suspected of abusing drugs or alcohol
7. Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Change in Sputum eosinophilia | At baseline and at the end of each of three dosing periods (every 16 weeks) for total study duration of 48 weeks.
  Absolute difference between the mean sputum eosinophil percent

SECONDARY OUTCOMES:
Change in Proportion of patients with sputum eosinophils ≤3% | At the start and end of each of three dosing periods (every 16 weeks) for total study duration of 48 weeks
  Number of patients with sputum eosinophils ≤3%
Change in Blood eosinophil count | At the start and end of each of three dosing periods (every 16 weeks) for total study duration of 48 weeks
  Absolute blood eosinophil count
Change in ACQ5 score | At the start and end of each of three dosing periods (every 16 weeks) for total study duration of 48 weeks
  Mean of 5-question Asthma Control Questionnaire
Change in FEV1 | At the start and end of each of three dosing periods (every 16 weeks) for total study duration of 48 weeks
  Forced expired volume in 1 second measured in litres
Change in Number of asthma exacerbations | At the start and end of each of three dosing periods (every 16 weeks) for total study duration of 48 weeks
  Number of asthma event that are defined as exacerbation (requiring increase in corticosteroids)
Change in Type of asthma exacerbations (as determined by quantitative sputum cytometry) | At the start and end of each of three dosing periods (every 16 weeks) for total study duration of 48 weeks
  Type of exacerbation shown by: neutrophilic, eosinophilic or mixed neutrophilic/eosinophilic bronchitis
Change in Proportion of patients requiring daily oral corticosteroid therapy | At the start and end of each of three dosing periods (every 16 weeks) for total study duration of 48 weeks
  Number of patients that require daily oral corticosteroids
Change in Cumulative systemic corticosteroid dose | At the start and end of each of three dosing periods (every 16 weeks) for total study duration of 48 weeks
  The total daily dose of oral corticosteroids

CONTACTS AND LOCATIONS:
Overall Officials: Parameswaran Nair, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- Firestone Institute of Respiratory Health, St Joseph's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mukherjee M, Lim HF, Thomas S, Miller D, Kjarsgaard M, Tan B, Sehmi R, Khalidi N, Nair P. Airway autoimmune responses in severe eosinophilic asthma following low-dose Mepolizumab therapy. Allergy Asthma Clin Immunol. 2017 Jan 6;13:2. doi: 10.1186/s13223-016-0174-5. eCollection 2017. PMID 28070196
- [Background] Mukherjee M, Forero DF, Tran S, Boulay ME, Bertrand M, Bhalla A, Cherukat J, Al-Hayyan H, Ayoub A, Revill SD, Javkar T, Radford K, Kjarsgaard M, Huang C, Dvorkin-Gheva A, Ask K, Olivenstein R, Dendukuri N, Lemiere C, Boulet LP, Martin JG, Nair P. Suboptimal treatment response to anti-IL-5 monoclonal antibodies in severe eosinophilic asthmatics with airway autoimmune phenomena. Eur Respir J. 2020 Oct 8;56(4):2000117. doi: 10.1183/13993003.00117-2020. Print 2020 Oct. PMID 32444405
- [Background] Mukherjee M, Bulir DC, Radford K, Kjarsgaard M, Huang CM, Jacobsen EA, Ochkur SI, Catuneanu A, Lamothe-Kipnes H, Mahony J, Lee JJ, Lacy P, Nair PK. Sputum autoantibodies in patients with severe eosinophilic asthma. J Allergy Clin Immunol. 2018 Apr;141(4):1269-1279. doi: 10.1016/j.jaci.2017.06.033. Epub 2017 Jul 24. PMID 28751233
- [Background] Passarell J, Jaworowicz D, Ludwig E, Rabinovich-Guilatt L, Cox DS, Levi M, Garin M, Fiedler-Kelly J, Bond M. Population Pharmacokinetic and Pharmacokinetic/Pharmacodynamic Modeling of Weight-Based Intravenous Reslizumab Dosing. J Clin Pharmacol. 2020 Aug;60(8):1039-1050. doi: 10.1002/jcph.1609. Epub 2020 Apr 25. PMID 32333684